CLINICAL TRIAL: NCT04472273
Title: Comparison of the Efficiency of High-Flow Nasal Cannula Oxygen Application and Classic Nasal Cannula Oxygen Application in Pediatric Patients With Sedation for Gastrointestinal System Endoscopy
Brief Title: Comparison of High-Flow Nasal Cannula Oxygen Application and Classic Nasal Cannula Oxygen Application
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kocaeli Derince Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Sami Olcay Özbay, MD, RESİDENT, Kocaeli Derince Education and Research Hospital
Other Study IDs: U1111-1253-6757
Record Dates: First submitted 2020-06-16; First posted 2020-07-15 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Sedation Complication
Keywords: high-flow oxygen therapy; pediatric outpatients; sedation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- high-flow nasal cannula group: Group 1
  Interventions: Procedure: high-flow nasal cannula / classic nasal cannula
- classic nasal cannula group: Group 2
  Interventions: Procedure: high-flow nasal cannula / classic nasal cannula

INTERVENTIONS:
Procedure: high-flow nasal cannula / classic nasal cannula — The oxygen given with nasal cannula cannot be humidified, causing drying in mucous membranes at high flow rates of more than 4L/min and problems in patient compliance.This situation prevents us to increase the oxygen FiO2 rate applied to the patient above 40%.According to the nasal cannula high-flow nasal cannula where heated and humidified oxygen can be delivered, oxygen therapy can be applied at a flow rate of 25L/min.It provides high flows easily, prevents the airway epithelium from drying out and improves mucus cleansing, causing a decrease in anatomical dead space.It provides discharge of expired air in the upper airways.It increases alveolar ventilation.It offers a stream adjusted to all children.Flow and titration can be adjusted according to the child's weight and effect.

SUMMARY:
Recently, sedation practices have increased for diagnostic and interventional procedures for children in non-operating rooms. On the other hand, the rate of respiratory complications especially in non-operating room sedation applications is quite high. Oxygen therapy in sedation applied to non-operating room endoscopy patients is mostly performed with classical nasal cannula. However, recently, the use of High-flow nasal cannula oxygen therapy has been increasing.

According to the classical nasal cannula oxygen therapy application where non-moistened oxygen is applied in high-flow nasal cannula oxygen therapy applications where heated and humidified oxygen can be delivered, oxygen therapy can be applied at a flow rate of 25L / min. This method has many advantages. Some of those; makes it possible to provide high flows easily, prevents the airway epithelium from drying out and improves mucus cleansing, causing a decrease in anatomical dead space. It provides discharge of expired air in the upper airways. It reduces the respiration of gas with high CO2 and decreased O2. It increases alveolar ventilation. It is easy to use and increases patient comfort. It offers a stream adjusted to all children. Flow and titration can be adjusted according to the child's weight and effect. Physiological evidence in the pediatric population indicates that flows equal to or higher than 2 L / kg / min produce clinically significant pharyngeal pressure, improve breathing and accelerate the emptying of the respiratory muscles. Because of all these features, high-flow nasal cannula oxygen therapy application is used safely in pediatric patients.

In general, it is reported that in non-operating room anesthesia, sedation or anesthesia applied in pediatric patients causes undesirable effects by 20%, most of them (5.5%) have respiratory complications and bradycardia due to hypoxemia.

In this study, we aimed to compare the respiratory and hemodynamic results of high-flow nasal cannula oxygen application, which is routinely used in sedation applications in the pediatric endoscopy unit of our hospital, with the classical nasal cannula oxygen therapy application.

DETAILED DESCRIPTION:
Recently, sedation practices have increased for diagnostic and interventional procedures for children in non-operating rooms. On the other hand, the rate of respiratory complications especially in non-operating room sedation applications is quite high. Oxygen therapy in sedation applied to non-operating room endoscopy patients is mostly performed with classical nasal cannula. However, recently, the use of High-flow nasal cannula oxygen therapy has been increasing.

Classical nasal cannula oxygen therapy application; It is a system made of plastic or rubber material with two open ends placed in the patient's nostrils. It is the most commonly used oxygen therapy application method. However, it has some disadvantages. The most important of these is that the oxygen given in this method cannot be humidified, causing drying in mucous membranes at high flow rates of more than 4 L / min and problems in patient compliance. This situation prevents us to increase the oxygen FiO2 rate applied to the patient above 40%.

According to the classical nasal cannula oxygen therapy application where non-moistened oxygen is applied in high-flow nasal cannula oxygen therapy applications where heated and humidified oxygen can be delivered, oxygen therapy can be applied at a flow rate of 25L / min. This method has many advantages. Some of those; makes it possible to provide high flows easily, prevents the airway epithelium from drying out and improves mucus cleansing, causing a decrease in anatomical dead space. It provides discharge of expired air in the upper airways. It reduces the respiration of gas with high CO2 and decreased O2. It increases alveolar ventilation. It is easy to use and increases patient comfort. It offers a stream adjusted to all children. Flow and titration can be adjusted according to the child's weight and effect. Physiological evidence in the pediatric population indicates that flows equal to or higher than 2 L / kg / min produce clinically significant pharyngeal pressure, improve breathing and accelerate the emptying of the respiratory muscles. Because of all these features, high-flow nasal cannula oxygen therapy application is used safely in pediatric patients.

In general, it is reported that in non-operating room anesthesia, sedation or anesthesia applied in pediatric patients causes undesirable effects by 20%, most of them (5.5%) have respiratory complications and bradycardia due to hypoxemia.

In this study, we aimed to compare the respiratory and hemodynamic results of high-flow nasal cannula oxygen application, which is routinely used in sedation applications in the pediatric endoscopy unit of our hospital, with the classical nasal cannula oxygen therapy application.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 4-18 years
* Patients undergoing gastroenterological intervention
* Patients undergoing sedation
* Patients with ASA 1-2 risk group
* Patients who have been informed of the study for informed consent

Exclusion Criteria:

* Patients under 4 years old and over 18 years old
* Patients with ASA 3 and above risk groups
* Patients who refuse to participate in the study

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children of 4-18 years of age, whose informed consent is signed by their parents.
Sampling Method: Non-Probability Sample
Enrollment: 82 (Estimated)
Dates: Start 2020-02-27 (Actual); Primary Completion 2020-10 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Comparison of the effects of high-flow nasal cannula oxygen administration and nasal cannula oxygen administration on respiratory parameters in patients undergoing sedation in the pediatric endoscopy unit. | SpO2 values of patients at admission, 1 minute, 5 minutes, 10 minutes, 15 minutes and 20 minutes will be recorded. After the procedure, SpO2 and ETCO2 values at the input, 1 minute, 5 minutes, 10 minutes, 15 minutes and 20 minutes will be recorded.
  SpO2 and ETCO2 are recorded as data in patients in high-flow nasal cannula and classical nasal cannula oxygen therapy applications.

SECONDARY OUTCOMES:
Comparison of the effects of high flow nasal cannula oxygen administration and nasal cannula oxygen administration on hemodynamic parameters in patients undergoing sedation in the pediatric endoscopy unit. | HR and blood pressure values of patients at admission, 1 minute, 5 minutes, 10 minutes 15 minutes and 20 minutes will be recorded. After the procedure, HR values at the input, 1 minute, 5 minutes, 10 minutes, 15 minutes and 20 minutes will be recorded.
  HR and blood pressure (both systolic and diastolic blood pressure) are recorded as data in patients in high-flow nasal cannula and classical nasal cannula oxygen therapy applications.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet YILMAZ, Study Director — Assistant Professor
Locations (1):
- Sami Olcay OZBAY, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided